CLINICAL TRIAL: NCT01251744
Title: Study of Maternal-foetal Cytomegalovirus (CMV) Transmission
Brief Title: Study of the Transmission of Cytomegalovirus (CMV) Infection From Mother to Foetus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113134
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-05

CONDITIONS: Infections, Cytomegalovirus; Cytomegalovirus Infections
Keywords: Pregnancy; Congenital; Cytomegalovirus infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection

ARMS (2):
- CMV Mothers' Group (Experimental): Pregnant subjects with confirmed primary CMV infection.
  Interventions: Procedure: Blood sample; Procedure: Cord blood sample; Procedure: Saliva swab; Procedure: Urine sampling; Procedure: Vaginal swab
- CMV Newborns' Group (Experimental): Offsprings of the CMV Mothers' Group, also tested for CMV infection, comprising infants that were live born.
  Interventions: Procedure: Blood sample; Procedure: Cord blood sample; Procedure: Saliva swab; Procedure: Urine sampling; Procedure: Vaginal swab

INTERVENTIONS:
Procedure: Blood sample — Blood sample at study entry, every two months during pregnancy, at pregnancy conclusion and one month after pregnancy conclusion.
Procedure: Cord blood sample — Cord blood sample taken at the time of delivery.
Procedure: Saliva swab — Saliva swab taken at study entry, every month during pregnancy, at pregnancy conclusion and one month after pregnancy conclusion.
Procedure: Urine sampling — Approximately 10 mL of urine will be sampled at study entry, every month during pregnancy, at pregnancy conclusion and one month after pregnancy conclusion.
Procedure: Vaginal swab — Vaginal swab taken at study entry, every month during pregnancy and one month after pregnancy conclusion.

SUMMARY:
This study is designed to evaluate maternal virological and immunological parameters to determine their ability to predict congenital cytomegalovirus (CMV) infection. When a pregnant woman is infected with CMV, her immune system (which protects her from infection) is activated and the virus can be found in the woman's bodily fluids (blood, saliva, urine, vaginal secretions). The aim of this study is to find out if there is a link between either the pregnant woman's immune response or the presence of the virus in these bodily fluids and the child/foetus being infected with the virus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol .
* A pregnant female, 18 years of age or older at the time of study enrolment.
* Women with confirmed primary CMV infection.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to study entry.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational pharmaceutical product.
* Previous vaccination against CMV infection.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history or physical examination
* Major congenital defects, serious chronic illness or organ transplantation.
* Administration of immunoglobulins and/or any blood products within the three months preceding study enrolment or during the pregnancy.
* Documented Human immunodeficiency virus (HIV)-positive subject.
* Gestational age of more than 34 weeks, as determined by foetal ultrasound.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-12-09 (Actual); Primary Completion 2013-11-06 (Actual); Study Completion 2015-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Belgium (7):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Mons
  - GSK Investigational Site, Wilrijk

REFERENCES:
- [Derived] Marchant A, Adali S, Alsdurf H, Bol V, Capelle X, De Schrevel N, Delroisse JM, Devlieger R, Dieussaert I, Donner C, Janssens M, Loquet P, Panackal AA, Seidl C, van den Berg RA, Paris R. Establishing Correlates of Maternal-Fetal Cytomegalovirus Transmission-One Step Closer Through Predictive Modeling. J Infect Dis. 2024 Dec 16;230(6):e1274-e1286. doi: 10.1093/infdis/jiae281. PMID 38865084
- [Derived] Antoine P, Olislagers V, Huygens A, Lecomte S, Liesnard C, Donner C, Marchant A. Functional exhaustion of CD4+ T lymphocytes during primary cytomegalovirus infection. J Immunol. 2012 Sep 1;189(5):2665-72. doi: 10.4049/jimmunol.1101165. Epub 2012 Aug 3. PMID 22865914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 82 pregnant subjects enrolled, 77 started this study: 4 were excluded from stat analyses; 1 had no available cytomegalovirus (CMV) infection status (IS) of her offsprings. Out of 82 offsprings, 78 newborns were enrolled (mothers signed informed consent) and 4 foetuses (stillbirth/termination) had CMV IS available but were not enrolled.
Groups:
- CMV Mothers' Group: Pregnant female subjects, 18 years of age or older at the time of study enrollment, with confirmed primary cytomegalovirus (CMV) infection.
Period: Overall Study
Arm/Group | CMV Mothers' Group | CMV Newborns' Group
Started | 77 | 78
Completed | 76 | 78
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CMV Mothers' Group | CMV Newborns' Group | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: This analysis presents data only for the CMV Mothers' Group.
  Years
    number analyzed (Participants) | 77 | 0 | 77
    (all) | 29.4 (4.8) |  | 29.4 (4.8)
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Population: This analysis presents data only for the CMV Newborns' Group.
  Weeks
    number analyzed (Participants) | 0 | 78 | 78
    (all) |  | 38.7 (2.5) | 38.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 42 | 119
  Male | 0 | 36 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic / North African Heritage | 3 | 2 | 5
  White - Caucasian / European Heritage | 74 | 71 | 145
  Unspecified | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Cytomegalovirus (CMV) Congenital Infection
Description: The CMV congenital infections were assessed in newborns and foetuses of subjects who had a confirmed primary CMV infection during pregnancy.
Time Frame: At Month 0
Population: The analysis was performed on the Total Enrolled cohort of Infant subjects, which included the newborns' group diagnosed with CMV infection and who had their medical records reviewed 1 month after birth and every 6 months for 2 years and foetus group, referring to infants that were stillborn or with pregnancy termination.
Measure: Count of Participants; unit: Participants
Groups:
- CMV Offsprings' Group: Offsprings of the CMV Mothers' Group, also tested for CMV infection.
- CMV Foetus Group: Offsprings of the CMV Mothers' Group, also tested for CMV infection, comprising infants that were stillborn or with pregnancy termination.
Arm/Group | CMV Offsprings' Group | CMV Newborns' Group | CMV Foetus Group
Number analyzed (Participants) | 82 | 78 | 4
Participants
  Confirmed CMV infection | 24 | 20 | 4
  Not confirmed CMV infection | 58 | 58 | 0

2. Primary Outcome: Number of Subjects With CMV Presence in the Urine
Description: Evidence of infection in urine was assessed by culture or by Polymerase Chain Reaction (PCR).
Time Frame: Within 10 days post-delivery (Days 0-9)
Population: The analysis was performed on the newborn sub-group in the Total Enrolled cohort of Infant subjects, which included the subjects diagnosed with CMV infection and who had their medical records reviewed 1 month after birth and every 6 months for 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Newborns' Group
Number analyzed (Participants) | 78
Participants
  Positive: PCR Not Done/Culture Positive | 6
  Positive: PCR Positive/Culture Negative | 5
  Positive: PCR Positive/Culture Not Done | 5
  Positive: PCR Positive/Culture Positive | 4
  Negative: PCR Negative/Culture Negative | 19
  Negative: PCR Negative/Culture Not Done | 6
  Negative: PCR Not Done/Culture Negative | 32
  Not Done: PCR Not Done/Culture Not Done | 1

3. Primary Outcome: Number of Subjects With CMV Presence in the Amniotic Fluid
Description: Evidence of infection in the amniotic fluid was assessed by culture or by Polymerase Chain Reaction (PCR).
Time Frame: Within 10 days post-delivery (Days 0-9)
Population: The analysis was performed on the Total Enrolled cohort of Infant subjects, which included the newborns sub-group diagnosed with CMV infection and who had their medical records reviewed 1 month after birth and every 6 months for 2 years and foetus sub-group, referring to infants that were stillborn or with pregnancy termination.
Measure: Count of Participants; unit: Participants
Groups:
- CMV Infant Group: Offspring of the CMV Mothers' Group, also tested for CMV infection.
- CMV Newborn Sub-Group: For the purpose of the analysis, this sub-group was divided from the CMV Infant Group, comprising infants that were live born.
- CMV Foetus Sub-Group: For the purpose of the analysis, this sub-group was divided from the CMV Infant Group, comprising infants that were stillborn or with pregnancy termination.
Arm/Group | CMV Infant Group | CMV Newborn Sub-Group | CMV Foetus Sub-Group
Number analyzed (Participants) | 82 | 78 | 4
Participants
  Positive: PCR Positive/Culture Negative | 9 | 7 | 2
  Positive: PCR Positive/Culture Positive | 6 | 4 | 2
  Negative: PCR Negative/Culture Negative | 28 | 28 | 0
  Negative: PCR Negative/Culture Not Done | 9 | 9 | 0
  Not Done: PCR Not Done/Culture Not Done | 30 | 30 | 0

4. Primary Outcome: Evidence of CMV DNA or CMV Inclusions in Tissues of an Aborted or Stillborn Foetus
Time Frame: Within 10 days post-delivery (Days 0-9)
Population: The diagnosis of CMV in the newborn was done according to the local standard of care and samples were not collected for this analysis.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

5. Primary Outcome: Number of CMV DNA Copies in Saliva, Urine, Blood or Vaginal Secretions
Description: The assessment focused on the presence of CMV DNA copies (by Quantitative Polymerase Chain Reaction [qPCR]) in saliva, urine, blood and vaginal secretions every month from study entry to, and including, pregnancy conclusion.
Time Frame: At Month 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort, which included all pregnant women with confirmed primary CMV infection and with available CMV infection status of the newborn, foetus or stillbirth.
Measure: Median (Inter-Quartile Range); unit: CMV DNA copies/sample
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
CMV DNA copies/sample
  Buffy coat | 0.000 [0.000 to 0.000]
  Plasma | 0.000 [0.000 to 0.000]
  Saliva | 0.000 [0.000 to 497.000]
  Urine | 1050.000 [0.000 to 3690.000]
  Vaginal mucus | 1950.000 [280.000 to 11510.00]

6. Primary Outcome: Number of CMV DNA Copies in Saliva, in Urine and in Blood or Vaginal Secretions
Description: The assessment focused on the presence of CMV DNA copies (by Quantitative Polymerase Chain Reaction [qPCR]) in saliva, urine and blood every month from study entry to, and including, pregnancy conclusion.
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: The analysis was performed on the Total Enrolled cohort, which included all pregnant subjects enrolled in this study, with available CMV infection status for their infants.
Measure: Median (Inter-Quartile Range); unit: CMV DNA copies/sample
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
CMV DNA copies/sample
  Buffy coat | 0.000 [0.000 to 0.000]
  Plasma | 0.000 [0.000 to 0.000]
  Saliva | 0.000 [0.000 to 231.500]
  Urine | 311.000 [0.000 to 1370.000]
  Vaginal mucus | 1950.000 [280.000 to 11510.00]

7. Primary Outcome: Descriptive Statistics of the Anti-CMV Immunoglobulin Type M (IgM) Status
Description: Anti-CMV IgM status was assessed by Enzyme-Linked Immunosorbent Assay [ELISA], with respect to positive and negative subjects. Grey Zone = optical density zone within 20% of cut-off value. When an optical density is within this grey zone, sample testing is repeated to confirm the result.
Time Frame: At Month 0
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 69
Participants
  Positive | 53
  Negative | 12
  Grey Zone | 4

8. Primary Outcome: Descriptive Statistics of the Anti-CMV IgM Status
Description: as for outcome 7
Time Frame: At Month 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 56
Participants
  Positive | 27
  Negative | 24
  Grey Zone | 5

9. Primary Outcome: Descriptive Statistics of the Anti-Cytomegalovirus (Anti-CMV) Immunoglobulin Type M (IgM) Status
Description: as for outcome 7
Time Frame: At Month 4
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 23
Participants
  Positive | 8
  Negative | 13
  Grey Zone | 2

10. Primary Outcome: Anti-CMV Immunoglobulin Type M (IgM) Status, Descriptive Statistics
Description: Anti-CMV IgM status was assessed by Enzyme-Linked Immunosorbent Assay [ELISA], with respect to positive and negative subjects.
Time Frame: At Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 4
Participants
  Positive | 1
  Negative | 3

11. Primary Outcome: Descriptive Statistics for the Anti-CMV IgM Status
Description: as for outcome 7
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 64
Participants
  Positive | 24
  Negative | 35
  Grey Zone | 5

12. Primary Outcome: Anti-glycoprotein B (gB) Immunoglobulin Type G (IgG) Antibody Concentrations
Description: Anti-gB IgG concentrations were assessed by ELISA, presented as geometric mean concentrations (GMCs) and expressed in ELISA units per milliliter (EU/mL). The cut-off value was greater than or equal to (≥) 54 EU/mL.
Time Frame: At Month 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort, which included all pregnant women with confirmed primary CMV infection, with available CMV infection status of the newborn, foetus or stillbirth and with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 69
EU/mL | 4460.8 [3432.2 to 5797.6]

13. Primary Outcome: Anti-gB IgG Antibody Concentrations
Description: as for outcome 12
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 64
EU/mL | 6708.2 [5835.9 to 7711.0]

14. Primary Outcome: Descriptive Statistics of the Anti-glycoprotein B (gB) Immunoglobulin Type G (IgG) Avidity Index
Description: The avidity index was calculated as the mean absorbance of reactions in which the immune complexes were exposed to urea divided by the mean absorbance of reactions in which the immune complexes were not exposed to urea, expressed as a percentage.
Time Frame: At Month 0
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 22.000 [17.000 to 35.000]

15. Primary Outcome: Descriptive Statistics of the Anti-gB IgG Avidity Index
Description: as for outcome 14
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 36.500 [28.000 to 43.000]

16. Primary Outcome: CMV-specific Cluster of Differentiation 4 (CD4) T-cell Frequencies
Description: Descriptive statistics of the frequency of CMV-specific CD4 T cells expressing at least two markers among: cluster of differentiation 40 ligand (CD40L), interleukin-2 (IL-2), interferon-gamma (IFN-γ), tumor necrosis factor-alpha (TNF-α), as assessed by Intracellular Cytokine Staining [ICS], by stimulating agent (among Human Cytomegalovirus [HCMV] immediate-early gene [IE1] antigen, HCMV glicoprotein B [gB] antigen, HCMV lysate antigen and HCMV pp65 antigen).
Time Frame: At Month 0
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: CMV-specific CD4 T cells/million T-cells
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 65
CMV-specific CD4 T cells/million T-cells
  HCMV IE1 Ag: number analyzed (Participants) | 64
  HCMV IE1 Ag | 350.50 [101.50 to 633.00]
  HCMV gB Ag: number analyzed (Participants) | 64
  HCMV gB Ag | 1009.50 [381.00 to 3395.00]
  HCMV lysate Ag: number analyzed (Participants) | 64
  HCMV lysate Ag | 2864.00 [1396.00 to 5980.00]
  HCMV pp65 Ag | 510.00 [258.00 to 813.00]

17. Primary Outcome: CMV-specific CD4 T-cell Frequencies
Description: Descriptive statistics of the frequency of CMV-specific CD4 T cells expressing at least two markers among CD40L, IL-2, IFNg, TNFa, as assessed by Intracellular Cytokine Staining [ICS], by stimulating agent (among immediate-early gene [IE1] antigen, glicoprotein B [gB] antigen, CMV lysate antigen and CMV pp65 antigen).
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: CMV-specific CD4 T cells/million T-cells
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 59
CMV-specific CD4 T cells/million T-cells
  HCMV IE1 Ag: number analyzed (Participants) | 58
  HCMV IE1 Ag | 261.00 [130.00 to 555.00]
  HCMV gB Ag | 830.00 [292.00 to 4407.00]
  HCMV lysate Ag: number analyzed (Participants) | 58
  HCMV lysate Ag | 2330.00 [1314.00 to 3724.00]
  HCMV pp65 Ag | 455.00 [236.00 to 761.00]

18. Primary Outcome: CMV-specific Cluster of Differentiation 8 (CD8) T-cell Frequencies
Description: Descriptive statistics of the frequency of CMV-specific CD8 T cells expressing at least two markers among CD40L, IL-2, IFNg, TNFa, as assessed by Intracellular Cytokine Staining [ICS], by stimulating agent (among immediate-early gene [IE1] antigen, glicoprotein B [gB] antigen, CMV lysate antigen and CMV pp65 antigen).
Time Frame: At Month 0
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: CMV-specific CD8 T cells/million Tcells
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 65
CMV-specific CD8 T cells/million Tcells
  HCMV IE1 Ag: number analyzed (Participants) | 64
  HCMV IE1 Ag | 1448.00 [496.50 to 7890.00]
  HCMV gB Ag: number analyzed (Participants) | 64
  HCMV gB Ag | 274.00 [88.00 to 770.50]
  HCMV lysate Ag: number analyzed (Participants) | 64
  HCMV lysate Ag | 30.50 [1.00 to 122.00]
  HCMV pp65 Ag | 1030.00 [243.00 to 2043.00]

19. Primary Outcome: CMV-specific CD8 T-cell Frequencies
Description: as for outcome 18
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: CMV-specific CD8 T cells/million T-cells
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 59
CMV-specific CD8 T cells/million T-cells
  HCMV IE1 Ag: number analyzed (Participants) | 58
  HCMV IE1 Ag | 2519.00 [548.00 to 9135.00]
  HCMV gB Ag | 209.00 [57.00 to 806.00]
  HCMV lysate Ag: number analyzed (Participants) | 58
  HCMV lysate Ag | 34.50 [1.0 to 122.00]
  HCMV pp65 Ag | 1054.00 [550.00 to 1931.00]

20. Primary Outcome: CMV-specific Proliferating Cluster of Differentiation (CD4) T Cells Frequencies
Description: Labelled cells were quantified by flow cytometry, by stimulating agent (among immediate-early gene [IE1] antigen, glicoprotein B [gB] antigen, CMV lysate antigen and CMV pp65 antigen).
Time Frame: At Month 0
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: CMV-specific CD4 Tcells/million T-cells
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 61
CMV-specific CD4 Tcells/million T-cells
  HCMV IE1 Ag: number analyzed (Participants) | 60
  HCMV IE1 Ag | -0.00 [-0.22 to 0.12]
  HCMV gB Ag: number analyzed (Participants) | 60
  HCMV gB Ag | 0.61 [0.21 to 1.33]
  HCMV lysate Ag: number analyzed (Participants) | 56
  HCMV lysate Ag | 4.37 [1.69 to 10.67]
  HCMV pp65 Ag | 0.07 [-0.09 to 0.26]

21. Primary Outcome: CMV-specific Proliferating CD4 T Cells Frequencies
Description: Labelled cells were quantified by flow cytometry, by stimulating agent (among immediate-early gene [IE1] antigen, glicoprotein B [gB] antigen, CMV lysate antigen and CMV pp65 antigen).
  Note: Results were retrieved by subtracting the background without imputing the negative and zero values, this generated negative values.
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: CMV-specific CD4 T cells/million T-cells
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 52
CMV-specific CD4 T cells/million T-cells
  HCMV IE1 Ag | -0.04 [-0.19 to 0.06]
  HCMV gB Ag | 0.53 [0.16 to 1.93]
  HCMV lysate Ag | 4.02 [2.49 to 13.43]
  HCMV pp65 Ag | 0.06 [-0.08 to 0.36]

22. Primary Outcome: Concentrations of Anti-CMV Tegument Protein Immunoglobulin G (IgG) Antibodies
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs), measured in units per milliliter (U/mL). Concentrations of antibodies were assessed by the Enzyme-Linked Immunosorbent Assay (ELISA) for a cut-off greater than or equal to (≥) 0.668 U/mL.
Time Frame: At Day 0 = study entry
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 69
U/mL | 4.8 [3.9 to 6.0]

23. Primary Outcome: Anti-CMV Tegument Protein Immunoglobulin G (IgG) Antibody Concentrations
Description: as for outcome 22
Time Frame: At Month 2
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 56
U/mL | 4.9 [3.8 to 6.5]

24. Primary Outcome: Concentrations of Anti-CMV Tegument Protein IgG Antibodies
Description: as for outcome 22
Time Frame: At Month 4
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 23
U/mL | 4.9 [3.2 to 7.5]

25. Primary Outcome: Anti-CMV Tegument Protein IgG Antibody Concentrations
Description: as for outcome 22
Time Frame: At Month 6
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 4
U/mL | 13.5 [3.9 to 46.2]

26. Primary Outcome: Concentrations of Anti-CMV IgG Antibodies
Description: as for outcome 22
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 64
U/mL | 5.3 [4.3 to 6.6]

27. Primary Outcome: Descriptive Statistics of the Anti-CMV Tegument Protein Globulin Type B (gB) Immunoglobulin G (IgG) Avidity, by Congenital Infection Status
Description: Avidity of anti-CMV tegument protein gB IgG was assessed by ELISA. The avidity index was calculated as the mean absorbance of reactions in which the immune complexes were exposed to urea divided by the mean absorbance of reactions in which the immune complexes were not exposed to urea, expressed as a percentage.
Time Frame: At Day 0 = study entry
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 23.000 [12.000 to 35.000]

28. Primary Outcome: Descriptive Statistics of the Anti-CMV Tegument Protein gB Immunoglobulin G (IgG) Avidity, by Congenital Infection Status
Description: as for outcome 27
Time Frame: At Month 2
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 24.500 [16.500 to 40.500]

29. Primary Outcome: Descriptive Statistics of the Anti-CMV Tegument Protein gB IgG Avidity, by Congenital Infection Status
Description: as for outcome 27
Time Frame: At Month 4
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 28.000 [22.000 to 44.500]

30. Primary Outcome: Descriptive Statistics of the Anti-CMV Tegument Protein Globulin Type B (gB) IgG Avidity, by Congenital Infection Status
Description: as for outcome 27
Time Frame: At Month 6
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 46.000 [29.500 to 50.500]

31. Primary Outcome: Anti-CMV Tegument Protein Globulin Type B (gB) Immunoglobulin G (IgG) Avidity Descriptive Statistics, by Congenital Infection Status
Description: as for outcome 27
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage (avidity index)
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 70
Percentage (avidity index) | 31.000 [18.000 to 44.000]

32. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Fibroblast)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 10 ED50.
Time Frame: At Month 0
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 68
titers | 282.5 [199.6 to 400.0]

33. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Fibroblast)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 10 ED50.
Time Frame: At Month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 56
titers | 456.9 [342.0 to 610.4]

34. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Fibroblast)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 10 ED50.
Time Frame: At Month 4
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 23
titers | 422.9 [308.1 to 580.7]

35. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Fibroblast)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 10 ED50.
Time Frame: At Month 6
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 4
titers | 550.3 [266.4 to 1136.8]

36. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Fibroblast)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 10 ED50.
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 64
titers | 583.9 [491.1 to 694.3]

37. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Epithelial Cells)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 15 ED50.
Time Frame: At Month 0
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 68
titers | 822.5 [642.5 to 1053.0]

38. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Epithelial Cells)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 15 ED50.
Time Frame: At Month 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 56
titers | 986.3 [746.2 to 1303.6]

39. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Epithelial Cells)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 15 ED50.
Time Frame: At Month 4
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 23
titers | 1147.6 [832.8 to 1581.4]

40. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Epithelial Cells)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 15 ED50.
Time Frame: At Month 6
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 4
titers | 2137.1 [675.4 to 6762.2]

41. Primary Outcome: Anti-CMV Antibody Titers, by Neutralisation Assay (Epithelial Cells)
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs), for the seropositivity cut-off of ≥ 10 ED50.
Time Frame: At pregnancy conclusion (Day 0 to 5, Day 0 = day of delivery, stillbirth or termination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CMV Mothers' Group
Number analyzed (Participants) | 64
titers | 1100.2 [898.8 to 1346.7]

ADVERSE EVENTS:
Time Frame: Serious adverse events were reported during the entire study period (From Day 0 to pregnancy conclusion).
Description: Only serious adverse events were collected in the study.
Arm/Group | CMV Mothers' Group | CMV Newborns' Group
All-Cause Mortality (participants affected / at risk) | 0/77 | 1/78
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/78
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMV Mothers' Group (N=77) | CMV Newborns' Group (N=78)
Death neonatal (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.